CLINICAL TRIAL: NCT03214614
Title: Assessment of Safety, Tolerability and Pharmacokinetics of Multiple Ascending Oral Doses of GLPG2451 and of the Combination of GLPG2451 and GLPG2222 in Healthy Male Subjects
Brief Title: A Study to Assess Safety, Tolerability and Pharmacokinetics of GLPG2451 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: GLPG2451-CL-105
Record Dates: First submitted 2017-07-10; First posted 2017-07-11 (Actual); Last update posted 2017-09-13 (Actual); Status verified 2017-09

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- GLPG2451 multiple dose (Experimental): Multiple doses of GLPG2451 oral suspension at up to 3 dose levels in ascending order
  Interventions: Drug: GLPG2451 multiple dose
- Placebo multiple dose (Placebo Comparator): Multiple doses of Placebo oral suspension
  Interventions: Drug: Placebo multiple dose
- GLPG2451/GLPG2222 (Experimental): Multiple doses of GLPG2451 oral suspension combined GLPG2222 oral suspension at up to 2 dose levels
  Interventions: Drug: GLPG2451/GLPG2222 multiple dose
- Combined Placebo multiple dose (Placebo Comparator): Multiple doses of Combined Placebo oral suspension
  Interventions: Drug: Combined Placebo multiple dose

INTERVENTIONS:
Drug: GLPG2451 multiple dose — GLPG2451 oral suspension, multiple ascending doses, daily for 14 days
  Arms: GLPG2451 multiple dose
Drug: Placebo multiple dose — Placebo, oral suspension, daily for 14 days
  Arms: Placebo multiple dose
Drug: GLPG2451/GLPG2222 multiple dose — GLPG2451 oral suspension and GLPG2222 oral suspension, multiple doses, daily for 14 days
  Arms: GLPG2451/GLPG2222
Drug: Combined Placebo multiple dose — Combined Placebo, oral suspension, daily for 14 days
  Arms: Combined Placebo multiple dose

SUMMARY:
The study is a Phase I, randomized, double-blind, placebo-controlled study evaluating multiple ascending oral doses of GLPG2451 and the combination of GLPG2451 and GLPG2222 given for 14 days in healthy male subjects.

The purpose of the study is to evaluate the safety and tolerability of multiple ascending oral doses of GLPG2451 given to healthy male subjects compared to placebo, as well as of multiple oral doses of the combination of GLPG2451/GLPG2222 compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male between 18 and 50 years of age inclusive, on the date of signing the Informed Consent Form (ICF).
* A body mass index (BMI) between 18-30 kg/m2, inclusive.
* Judged by the investigator to be in good health based upon the results of a medical history, physical examination, vital signs, 12-lead ECG, and clinical safety laboratory tests prior to the initial study drug administration. Clinical safety laboratory test results must be within the laboratory reference ranges or test results that are outside the reference ranges need to be considered non clinically significant in the opinion of the investigator. One retest is allowed during screening period, if deemed appropriate by the investigator.
* Liver function tests must meet the following criteria: a. Aspartate aminotransferase (AST), ALT, or alkaline phosphatase (ALP) <1.5x ULN.

  b. Bilirubin not greater than ULN, however documented Gilbert's syndrome is acceptable but no more than one subject with confirmed Gilbert's syndrome is allowed per cohort. One retest is allowed during screening period, if deemed appropriate by the investigator.
* Able and willing to comply with restrictions on prior and concomitant medication as described in the protocol.
* Non-smokers and non-users of any nicotine-containing products. A non-smoker is defined as an individual who has abstained from smoking for at least 1 year prior to screening. A non-user is defined as an individual who has abstained from any nicotine containing products for at least 1 year prior to the screening.
* Negative urine screen for drugs of abuse (amphetamines, barbiturates, benzodiazepines, cannabis, cocaine, opiates, methadone, and tricyclic antidepressants) and negative alcohol breath test.
* No evidence of lens opacity on slit lamp examination or similar system (e.g. ITrace technology).
* Agree to the use of a highly effective method of contraception (see protocol).
* Able and willing to sign the ICF as approved by the IEC, prior to any screening evaluations and willing to adhere to predefined prohibitions and restrictions.

Exclusion Criteria:

* Known hypersensitivity to study drug ingredients or a significant allergic reaction to any drug as determined by the investigator, such as anaphylaxis requiring hospitalization.
* Positive serology for hepatitis B virus surface antigen (HBs Ag), hepatitis C virus (HCV), or history of hepatitis from any cause with the exception of hepatitis A.
* History of or a current immunosuppressive condition (e.g., human immunodeficiency virus [HIV] infection).
* Clinically significant illness in the 3 months before the initial study drug administration.
* Presence or sequelae of gastrointestinal, liver, kidney (creatinine clearance ≤80 mL/min using the Cockcroft-Gault formula; if calculated result ≤80 mL/min, a 24-hour urine collection to determine actual value can be performed) or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of drugs.
* History of malignancy within the past 5 years (except for basal cell carcinoma of the skin that has been treated and with no evidence of recurrence).
* Treatment with any drug known to have a well-defined potential for toxicity to a major organ in the last 3 months of 5 half-lives of the drug (whichever is the longer) before the initial study drug administration.
* Active drug or alcohol abuse (more than 3 glasses of wine or beer or equivalent/day) within 2 years prior to the initial study drug administration.
* Participation in a drug, drug-device combination or biologic investigational research study within 12 weeks or 5 half-lives of the investigational drug (whichever is the longer) prior to initial study drug administration.
* Any condition or circumstances that in the opinion of the investigator may make a subject unlikely or unable to complete the study or comply with study procedures and requirements.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 39 (Actual)
Dates: Start 2016-11-14 (Actual); Primary Completion 2017-08-25 (Actual); Study Completion 2017-08-25 (Actual)

PRIMARY OUTCOMES:
Change versus placebo in the proportion of subjects with adverse events | Between screening and 154 days after the last dose
  To assess safety and tolerability of multiple ascending doses and combination of GLPG2451 with GLPG2222 versus placebo in healthy subjects

SECONDARY OUTCOMES:
Maximum observed plasma concentration of GLPG2451 (Cmax) given alone or in combination with GLPG2222 | Between screening and 154 days after the last dose
  To characterize the pharmacokinetics of GLPG2451 and its metabolite after multiple oral doses in healthy subjects
Time of occurrence of Cmax for GLPG2451 given alone or in combination with GLPG2222 | Between screening and 154 days after the last dose
  To characterize the pharmacokinetics of GLPG2451and its metabolite after multiple oral doses in healthy subjects
Area under the plasma concentration-time curve of GLPG2451 (AUC0-t) given alone or in combination with GLPG2222 | Between screening and 154 days after the last dose
  To characterize the pharmacokinetics of GLPG2451 and its metabolite after multiple oral doses in healthy subjects
Ratio of 4-beta-hydroxycholesterol/cholesterol in plasma after multiple oral doses in healthy subjects | Day 1 predose and Day 14
  To explore the potential of CYP3A4 interaction with GLPG2451

CONTACTS AND LOCATIONS:
Overall Officials: Chris Brearley, MD, Study Director — Galapagos NV
Locations (1):
- SGS LSS Clinical Pharmacology Unit Antwerp, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: Undecided